CLINICAL TRIAL: NCT01617720
Title: MITRAFIT Cardinal Adjustable Mitral Repair Follow-up International Postmarketing Surveillance (PMS)
Brief Title: MITRAFIT- Cardinal Adjustable Mitral Repair Follow-up International Postmarketing Surveillance (PMS)
Acronym: MITRAFIT
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: VC1-2
Record Dates: First submitted 2012-06-07; First posted 2012-06-12 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Mitral Regurgitation
Keywords: mitral; valve; annuloplasty; mitral regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This Study is designed to observe the clinical outcomes of patients requiring mitral repair that were treated with the CE certified Cardinal System.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient is a candidate for mitral valve repair, with our without concomitant procedures.
* Subject is willing to give informed consent for collection of his/her clinical data.

Exclusion Criteria:

* Severe organic lesions with retracted chordae
* Congenital malformations with lack of valvular tissue
* Severe valvular calcifications
* Evolving bacterial endocarditis
* Known Sensitivity to Nickel or Chromium

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are candidate for mitral valve repair, with our without concomitant procedures.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2012-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
• Ability of the Cardinal ring to reduce mitral valve regurgitation | 30 day
• Percentage of patients in whom the size of the ring is adjusted | 6 months
• Technical feasibility of adjustment. | 6 months
  The ability of the surgeon to adjust the Cardinal ring when required, will be measured on a scale of 1-3 (1- successfull, 3- unsuccessful)
• The occurrence of serious device related adverse events in all patients. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ottavio Alfieri, Prof, MD, Principal Investigator — Hospital San Raffaele, Milan, Italy; Nicolas Doll, Prof, MD, Principal Investigator — SANA Herzchirurgie Stuttgart , Germany; Ehud Raanani, Prof, MD, Principal Investigator — Sheba Medical Center; Patrik Nataf, Prof, MD, Principal Investigator — Bichat Hospital; Volkmar Falk, Prof, MD, Principal Investigator — Zurich University, Zurich, Switzerland
Locations (2):
- SANA Herzchirurgie, Stuttgart, Germany
- Hospital San Rafaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.

REFERENCES:
- [Background] Sundermann SH, Czesla M, Kempfert J, Walther T, Nataf P, Raanani E, Jacobs S, Alfieri O, Maisano F, Falk V. Results of mitral valve repair with an adjustable annuloplasty ring 2 years after implantation. Heart Vessels. 2017 Jul;32(7):843-849. doi: 10.1007/s00380-016-0934-7. Epub 2016 Dec 23. PMID 28012074